CLINICAL TRIAL: NCT06491186
Title: Femoral Artery Ultrasound With Compressibility Assessment as a Method for Pulse Checks in Out-of-Hospital Cardiac Arrest: A Prospective Exploratory Study.
Brief Title: Pulse Checks Using Femoral Artery B-Mode Ultrasound With Compressibility Assessment
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Ludwig Boltzmann Institute Digital Health and Patient Safety (Other); Emergency Medical Service of Vienna (Unknown)
Responsible Party: Principal Investigator, Philipp Metelka, Resident, Medical University of Vienna
Other Study IDs: 1236/2024
Record Dates: First submitted 2024-05-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Cardiac Arrest; Out-of-hospital Cardiac Arrest; OHCA; Ultrasound; Point-Of-Care Ultrasound; POCUS; Pulse Check; POCUS Pulse Check; B-mode Ultrasound; Femoral Artery; Arterial Compressibility Assessment
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients
  Interventions: Other: Point of Care Ultrasound

INTERVENTIONS:
Other: Point of Care Ultrasound — Point-of-care ultrasound will be used to image the femoral vessels and to assess the presence or absence of a pulse and the compressibility of the artery during rhythm checks.

SUMMARY:
The goal of this prospective observational study is to investigate B-mode point-of care ultrasound with arterial compressibility assessment on the femoral artery as a method to determine the presence of a pulse and to compare it with concurrently conducted manual pulse checks.

DETAILED DESCRIPTION:
In this prospective observational study, a dedicated research team will be dispatched to cardiac arrest patients treated in the prehospital environment by emergency medical services (EMS). The team will use a portable ultrasound device to identify the femoral artery and employ B-mode ultrasound during rhythm checks. These ultrasound pulse checks will be conducted in parallel with the normal treatment of the patient, including manual pulse checks, and will only be conducted if ultrasound is possible without interference in the resuscitation. All treatment decisions will rest with the treating EMS team.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest treated by EMS
* Minimum age of 18 years

Exclusion Criteria:

* Pregnancy or suspected pregnancy
* Disapproval of the treating EMS team
* Adults under legal guardianship
* Inability to perform femoral artery doppler ultrasound due to limited access to the patient and possible interference with the treating EMS team
* Inability to perform femoral artery doppler ultrasound due to injuries or anatomic abnormalities in the femoral region or necessary emergent medical interventions in the femoral region
* Decision to transfer the patient to the hospital with ongoing CPR for emergent procedures such as extracorporeal CPR before femoral artery doppler ultrasound could be attempted
* Inability to safely perform femoral artery doppler ultrasound due to environmental hazards

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises non-pregnant adults suffering out-of-hospital cardiac arrest of any cause who are treated with CPR by emergency medical services.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Results of POCUS pulse check | During cardiac arrest, up to 45 minutes
  If the femoral artery is both non-compressible and pulsatile, the POCUS pulse check will be considered positive
Results of the concurrently conducted manual pulse check | During cardiac arrest, up to 45 minutes
  Parallel to our study team the treating team will conduct standard care, consisting of determining the presence or absence of a pulse by palpation. The results of these manual pulse checks will be recorded by our study team.

SECONDARY OUTCOMES:
Arterial compressibility during chest compressions | During cardiac arrest, up to 45 minutes
  Before each pulse check, during the last 30 seconds of cardiac compressions, the research team will apply pressure with the ultrasound probe until complete collapse of the femoral vein and visually assess if the neighbouring femoral is compressible as well.
Arterial compressibility during rhythm checks | During cardiac arrest, up to 45 minutes
  The compressibility of the femoral artery during rhythm checks (part of the "POCUS pulse check" primary outcome) will be recorded and analysed, independently of pulsatility
Arterial pulsatility during rhythm checks | During cardiac arrest, up to 45 minutes
  The pulsatility of the femoral artery during rhythm checks (part of the "POCUS pulse check" primary outcome) will be recorded and analysed, independently of compressibility
Time needed for POCUS pulse checks | During cardiac arrest, up to 45 minutes
  The POCUS pulse checks will be recorded and the time until presence or absence of a pulse could be determined will be recorded in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Metelka, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Emergency Medical Service of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided